CLINICAL TRIAL: NCT06651203
Title: Evaluation of the KIR3DL2 Marker in Flow Cytometry for Sézary Syndrome Diagnosis, Therapeutic Response and Residual Disease: a Prospective and Multicenter Study
Acronym: KISS01
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220915
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Mycosis Fungoides/Sezary Syndrome; Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, punch skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with clinical features consistent with erythrodermic cutaneous T cell lymphoma (CTCL): at initial diagnosis assessment
  Interventions: Other: Follow-up
- Patients previously diagnosed with Sézary syndrome (SS) and followed at Saint-Louis hospital

INTERVENTIONS:
Other: Follow-up — Clinical evaluation Blood sample Skin biopsy
  Groups: Patients with clinical features consistent with erythrodermic cutaneous T cell lymphoma (CTCL)

SUMMARY:
Cutaneous T-cell lymphomas (CTCL) are a group of primary cutaneous lymphomas including Mycosis Fungoides (MF) and Sézary syndrome (SS). SS is characterized by erythroderma and high numbers of circulating atypical lymphocytes (Sézary cells. SCs). Blood staging was added to the Tumor Node Metastasis (TNM) classification of MF/SS, reflecting the broad spectrum of CTCLs and the poor prognosis related to blood involvement. Blood classes were defined using blood-smear manual counts. However, this method never reached an international consensus status because of its subjective nature and its poor sensitivity. Several markers have been identified with variable efficiency for MF/SS diagnosis, outcome prediction and blood response to treatment. Such markers are essential for sharing and publishing consistent data about diagnosis, staging, prognosis and response to therapies. The detection of SCs is based on the lack of pan T-cell markers such as CD7 and/or CD26, which is not constant and may be observed in benign dermatoses. Thus, patients are often diagnosed with a delay, even treated with inappropriate therapies which worsens their prognosis. The relevance of blood-class in MF/SS is not only related to stage but also contributes to the response to therapy in clinical trials. We found that a significant proportion of benign T-cells from SS patients are CD4+CD26-, which may underestimate the rate of complete response to treatment. The identification of KIR3DL2 on SCs by our team has greatly helped the detailed study of the malignant clone. We have recently published two ancillary studies demonstrating the specificity and reliability of KIR3DL2 as a positive marker for SCs, and its prognosis value at initial diagnosis. We have designed an optimized flow-cytometry strategy as part of the routine care of erythrodermic patients at Saint-Louis Hospital and published in 2019 the results of a 5 years prospective single-center study involving 254 CTCL patients at initial diagnosis. We provided recommendations with the use a threshold value of KIR3DL2+SCs ≥ 200/µL or KIR3DL2+SCs/lymphocytes ≥ 10% in the diagnostic criteria and proposed a novel algorithm blood staging.

Several innovative immunotherapies in phase I/II trials or under compassionate use are ongoing in French centers, with the need to assess blood response using positive markers. Our goal is to validate KIR3DL2 as a specific marker for SS and to assess its reliability for blood staging and response to treatment in a multicenter study (11 centers).

ELIGIBILITY:
Inclusion criteria for all patient :

* Age ≥ 18
* Patients with health insurance
* Patients informed and not opposed to the study

Inclusion criteria for group 1 :

- Patients with clinical features consistent with erythrodermic CTCL at initial diagnosis.

Inclusion criteria for group 2 :

* Confirmed SS (previously diagnosed), followed at Saint Louis hospital participating center with all the following criteria:

  1. Stage T4 erythroderma (stage (erythrodermia ≥ 80% of total body area)
  2. The presence of an identical T-cell clone evidenced in blood and skin
  3. B2 blood staging at initial diagnosis

     Exclusion Criteria:
* Other progressive neoplastic disease
* Progressive psychotic disease
* Patient under guardianship or curatorship
* Patients with state medical aid
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with clinical features consistent with erythrodermic CTCL upon initial diagnosis assessment
  2. Patients previously diagnosed with SS and followed at Saint-Louis hospital
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of KIR3DL2 in the diagnosis of Sezary syndrome | At baseline, for group 1
  Defined as the proportion of patients KIR3DL2 <200/mm3 among patients without SS.
  Diagnosis of SS is defined as the presence of each of the following criteria:
  * T4 tumoral stage (erythrodermia ≥ 80% of total body area)
  * the presence of an identical T-cell clone evidenced in blood and skin
  * B2 blood stage
  Of note, according to ISCL/EORTC recommendations, FCM (Flow cytometry) blood staging is defined as:
  Stage B2: Expanded CD4+T cells with either CD4+CD26-≥30%, or CD4+CD7-≥40% And/or either CD4+CD7- or CD4+CD26-Tcells≥1000/mm3
  Stage B1: Either CD4+CD7- or CD4+CD26-T-cells ≥250/mm3, but not meeting B2 criteria
  Stage B0: CD4+CD7- and CD4+CD26-T-cells<250/mm3
  Diagnosis and KIR3DL2 measurements will be performed using standardized/harmonized procedures across participating laboratories, using the same combination of labelled antibodies, gating strategies and instrument settings.

SECONDARY OUTCOMES:
Receiver Operating Characteristics (ROC) curve (Sensitivity, Specificity, area under the ROC curve) of KIR3DL2 in the diagnosis of SS and mycosis fungoides (MF) in eligible patients. | At baseline, for group 1
  The reference diagnosis of SS will be defined as in the primary endpoint. KIR3DL2 will be measured with by FCM. Sensitivity, Specificity and ROC curve will be estimated both with the absolute count of KIR3DL2 and with the percentage of KIR3DL2 within lymphocyte subset.
Positive and Negative predictive values of KIR3DL2 for SS diagnosis in the population of patients with clinical features consistent with erythrodermic CTCL | Up to 24 months for group 1 patients
  Cut-off value used for KIR3DL2 : 200/mm3
Blood response | At 3 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 6 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 9 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 12 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 15 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 18 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 21 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Blood response | At 24 months for group 1 and 2
  Blood response using FCM and CD7 and CD26 markers as per latest ISCL and EORTC guidelines, with the definition of:
  Complete response (CR) : B0 stage. Partial response (PR) : > 50% decrease in quantitative measurements of blood tumor burden from baseline in those with B2 stage at baseline.
  Progressive disease (PD) : B0 to B2 or >50% increase from baseline and at least 5000 neoplastic cells/ mm3 or Loss of response: in those with PR who were originally B2 at baseline, > 50% increase from nadir. Stable disease (SD) : Fails to attain criteria for CR, PR, or PD. Relapse : increase of neoplastic blood lymphocytes to ≥ B2 in those with CR.
Overall survival | Up to 24 months for group 1
Progression free survival | Up to 24 months for group 1
Minimal Residual Disease | At 24 months for group 1 and 2
  Minimal Residual Disease (MRD) by multiparameter flow cytometric immunophenotyping and High Throughput Sequencing (HTS) based detection of clonal TCR gene rearrangements in patients with SS, at the time of CR remission, in comparison with baseline measurements on frozen PBMC.
Evolution to SS diagnosis as defined in the primary endpoint in stage B1 patients with KIR3DL2≥ 200/mm3 or ≥ 10% at baseline | Up to 24 months for group 1

IPD SHARING:
Plan to Share IPD: Undecided